CLINICAL TRIAL: NCT05686148
Title: The Effect of Vibration Application on Pain and Satisfaction Associated With Subcutaneous Anticoagulation Injection: A Randomized Crossover Study
Brief Title: The Effect of Vibration Application on Pain and Satisfaction Associated With Subcutaneous Anticoagulation Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, DİLEK YILDIRIM, Assistant Prof., Istanbul Aydın University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Vibration Subcutaneous inj
Record Dates: First submitted 2022-12-30; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Pain
Keywords: Acute Pain; Personal Satisfaction; Injections, Subcutaneous
MeSH Terms: conditions — Pain; Acute Pain; Personal Satisfaction | interventions — Vibration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All of the outcomes results were obtained by another researcher blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Vibration will be applied to the injection site for 5 minutes before the procedure.
  Interventions: Other: Vibration
- Control (No Intervention): No application will be made

INTERVENTIONS:
Other: Vibration — The device used for vibration application is produced to control pain and direct attention by providing 6000/min vibration. According to Melzack and Wall's Gate Control Theory, the application of local vibration reduces perceived pain by stimulating nerve fibers. Therefore, it should be ensured that the device is in full contact with the skin. The device can be used again by wiping with 70% alcohol. The device is placed 3 cm above the area to be injected. Vibration is applied to the area for 5 minutes before the procedure.
  Arms: Intervention

SUMMARY:
This study was needed to relieve the pain associated with subcutaneous injection, which is an application performed by nurses, to increase patient satisfaction, to increase patient compliance with treatment, and to strengthen positive patient-nurse communication.

The purpose of this study is to assess the effect of vibration stimulation application on subcutan injection induced pain and patient satisfaction. The study will be carried out in the internal medicine service of a university hospital. Vibration will be applied during subcutaneous injection of anticoagulant to one group, but not to the other group. It was planned to include 85 patients in the study.

DETAILED DESCRIPTION:
This study was needed to relieve the pain associated with subcutaneous injection, which is an application performed by nurses, to increase patient satisfaction, to increase patient compliance with treatment, and to strengthen positive patient-nurse communication.

The purpose of this study is to assess the effect of vibration stimulation application on subcutan injection induced pain and patient satisfaction.

The study will be conducted between September 2022 and January 2023 in the internal medicine ward of a university hospital in Istanbul/Turkey in a prospective, randomized, single-blind, crossover design.Two groups will be formed according to the crossover order. Volunteers will be informed about the study and their written consent will be obtained. Patient evaluation form, visual pain form and satisfaction scale will be applied to all patients before injection. The height, weight and body mass index of the patients will be measured by the specialist nurse. An anticoagulant will be administered subcutaneously over the abdominal region. The areas to be injected will be determined in the same way for each patient. Low molecular weight heparin will be administered subcutaneously to the umbilical region with and without vibration, with an interval of 24 hours. All patients will be injected with the same investigative nurse, following the standard procedure. 5 minutes after the application, the pain and satisfaction level of all patients will be evaluated using scales. Vibration application will be applied by the researchers for 5 minutes before the injection application.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers aged 18 and over,
* are conscious and have no communication problems,
* body mass index (BMI) of 18.5 to 30kg/m2,
* who have not had an injection in the last two weeks in the area to be injected subcutaneously,
* no signs of skin pain, hematoma, necrosis, scarring, incision or infection at the subcutaneous injection site,
* patients treated with subcutaneous heparin injection therapy

Exclusion Criteria:

* patients not receiving heparin injection therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-01-15 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Patient Information Form | day 1
  It includes some socio-demographic characteristics of the individual (age, gender, place of residence, marital status, educational status, employment status).
Visual Analog Scale | day 1
  Scale, 10 cm long, horizontal or vertical; It consists of a line starting with "No Pain" and ending with "Unbearable Pain". The use of VAS should be explained to the patient very well. The patient is asked to indicate the severity of the pain with a sign on this line where he deems appropriate. The distance between the onset of no pain and this point is measured in cm and recorded. Values range from 0 to 10, and patients' pain levels are evaluated over 10 points as 0 = no pain, 10 = unbearable pain.
Visual Analog Scale | day 2
  Scale, 10 cm long, horizontal or vertical; It consists of a line starting with "No Pain" and ending with "Unbearable Pain". The use of VAS should be explained to the patient very well. The patient is asked to indicate the severity of the pain with a sign on this line where he deems appropriate. The distance between the onset of no pain and this point is measured in cm and recorded. Values range from 0 to 10, and patients' pain levels are evaluated over 10 points as 0 = no pain, 10 = unbearable pain.
Visual Patient Satisfaction Scale | day 1
  The visual patient satisfaction scale combines with the features of the well-known VAS (Visual Analogue Scale). It consists of a 100 mm horizontal line without numbers. At one end of the line is the phrase "I am not satisfied at all" and at the other end is the statement "Very satisfied". The patient must synthesize all the components that affect him in relation to the medical care given, determine the state of satisfaction he is in and find the point on the line that corresponds to his situation.
Visual Patient Satisfaction Scale | day 2
  The visual patient satisfaction scale combines with the features of the well-known VAS (Visual Analogue Scale). It consists of a 100 mm horizontal line without numbers. At one end of the line is the phrase "I am not satisfied at all" and at the other end is the statement "Very satisfied". The patient must synthesize all the components that affect him in relation to the medical care given, determine the state of satisfaction he is in and find the point on the line that corresponds to his situation.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydin University, Istanbul, Turkey (Türkiye)